CLINICAL TRIAL: NCT02989207
Title: Comparing Surgical Approaches to Treat Black African and Africa-Caribbean Patients With Uncontrolled Primary Open Angle Glaucoma: A Randomised Feasibility Study
Brief Title: Surgical Approaches in Treating Uncontrolled Glaucoma in Black African and African-Caribbeans
Acronym: PEACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 160807; 15/LO/1810 (Other: Health Reseach Authority)
Record Dates: First submitted 2016-12-02; First posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Glaucoma; Trabeculectomy; Glaucoma drainage implant; Africa and Africa-Caribbean
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Trabeculectomy; Mitomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Trabeculectomy with Mitomycin-C (Active Comparator): The current standard surgical treatment for glaucoma remains trabeculectomy.
  Interventions: Procedure: Trabeculectomy; Drug: mitomycin-C
- Baerveldt tube surgery with Mitomycin C (Active Comparator): It consists of a tube, draining aqueous humour to a plate
  Interventions: Device: Baerveldt tube surgery; Drug: mitomycin-C
- Baerveldt tube surgery without Mitomycin C (Active Comparator): It consists of a tube, draining aqueous humour to a plate
  Interventions: Device: Baerveldt tube surgery

INTERVENTIONS:
Procedure: Trabeculectomy — The current standard surgical treatment for glaucoma remains trabeculectomy. Wound healing modulation with antifibrotic agents, like MMC and 5-fluorouracil (5-FU), has been shown to increase the success of glaucoma filtering surgery in high-risk eyes
  Other Names: Trabeculectomy with Mitomycin-C
  Arms: Trabeculectomy with Mitomycin-C
Device: Baerveldt tube surgery — All glaucoma drainage devices consist of a tube which is inserted into the anterior chamber of the eye, draining aqueous humour to a plate which maintains a minimum bleb size and allows the collection of aqueous humour to be absorbed into the surrounding tissue.
  Other Names: Baerveldt tube surgery with Mitomycin C
  Arms: Baerveldt tube surgery with Mitomycin C; Baerveldt tube surgery without Mitomycin C
Drug: mitomycin-C — This is an anti scarring agent whcih is an standard adjunctive treatment in glaucoma surgery
  Arms: Baerveldt tube surgery with Mitomycin C; Trabeculectomy with Mitomycin-C

SUMMARY:
The aim is to perform a randomised feasibility trial preceding a large prospective randomised controlled trial (RCT) comparing three surgical methods - trabeculectomy with Mitomycin C (MMC), primary Baerveldt tube with MMC and Baerveldt tube without MMC - in black African/African Caribbean patients with Primary Open Angle Glaucoma (POAG) living in London.

The UK Office of National Statistics estimated that among the population of England in 2007, approximately 4.3% were of African/African-Caribbean background, while in large cities such as London and Birmingham about 20% of the population is of African/African-Caribbean origin. For eye units in these cities, managing glaucoma in this population is challenging and we need to identify a better alternative to our current standard surgical treatment.

There is now evidence from one RCT which shows better overall outcomes from tube surgery in comparison to trabeculectomy for glaucoma. However, this study did not address black populations specifically and did not address the potential role of MMC in tube surgery.

This feasibility study will enable us to design a fully powered RCT with the aim of determining how best to optimise the surgical treatment of POAG in black populations, by comparing outcomes in three types of glaucoma surgery.

DETAILED DESCRIPTION:
An audit performed at St Thomas's Hospital in 2008 showed that 52 trabeculectomy and 50 Baerveldt tube procedures were done in one year, with 60% of the patients being of 'black' ethnicity. This audit provides the basis for teh recruitment target. Assuming that the majority of the trabeculectomies performed were for POAG then most of these 'black' patients would have been eligible for the trial.

Primary Tube versus Trabeculectomy Study (PTVT) St Thomas' Hospital is the leading recruiting centre for this multinational study. The investigators have recruited over 50 patients in the last 2 years despite the lack of a dedicated research team. The trial retention rate has also been very good with less than 5% loss to follow-up rates.

Patient Feedback and Involvement The proposed research was reviewed in a feedback session in 2012 with 5 black African-Caribbean/African patients with glaucoma attending St Thomas' Hospital. All were very positive about the potential trial and all understood that there is a 'unique' problem for glaucoma surgery in this group of patients. Suggestions for the trial included more emphasis on the importance of treatment for glaucoma, disseminating information about the trial in community centres, and the possibility of expert patients who can act as patient advocates and help with recruitment in the glaucoma clinics and present the study in local community centres.

Feasibility study This protocol is for a randomised feasibility trial which will compare standard treatment (trabeculectomy with MMC) with primary Baerveldt tube surgery with or without MMC in black African/African-Caribbean patients with POAG living in London. The study will look at the feasibility of recruitment for a proposed larger scale RCT and will also help the investigators to refine the methodology for the proposed trial in terms of outcome measures and analysis. It will also help the investigators to recruit a patient user group for input into the conduct and monitoring of the main trial.

Information the study will provide

The investigators are conducting this feasibility study in order to get an estimate of the likely recruitment rate for the main study and to collect information that will help the investigators to refine the outcome measures for the main study and to allow a valid calculation of the sample size needed for a definitive study to answer the primary research question. The investigators will use questionnaires to gather data on patients' quality of life for health economic analysis but it is also our hope that the questionnaires will give the investigators information on the perspectives of patients, including their preferences. This feasibility study will help the investigators to explore how they can gather useful information on the patient perspective.

The feasibility study will also inform their planning for the main trial and data management and help them to develop their community engagement and recruitment strategies, including theri strategy for publicising the trial and enhancing recruitment. In addition, the investigators intend to use the feasibility study to recruit a patient representative group for input into the conduct and monitoring of the proposed main study.

Risks and benefits The potential risks and benefits for patients participating in the feasibility study are similar to those for standard clinical care. All participants will have been identified as in need of glaucoma drainage surgery. Both trabeculectomy (currently as first line treatment) and Baerveldt tube surgery (currently as second line treatment) are in routine use for the treatment of POAG. Evidence on the beneficial effect of MMC is equivocal. First line treatment with Baerveldt tube surgery may be associated with less failure and complications than first line treatment by trabeculectomy but there is as yet no definitive evidence on this question that is specific to the population included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the information sheet and give informed consent.
* Black African Caribbean or African (defined as a person having origins in any of the black racial groups of Africa). The identification of African or African-Caribbean ethnicity will be based on patients' self-reported ethnicity classification in their NHS case notes. In our recent audit, almost 90% of the case notes had data on patients' self-reported ethnicity.
* Age 18 to 85 years, inclusive. Inclusion criteria for study eye

All of the criteria listed below must be present in the study eye in order for the patient to be eligible for enrolment in the study:

• Glaucoma that is uncontrolled on tolerated medical therapy with IOP ≥18 mmHg and ≤40 mmHg in the study eye.

• No previous incisional ocular surgery in the study eye except for: i) Clear corneal phacoemulsification surgery. ii) Previous conjunctival sparing minimally invasive glaucoma surgeries (MIGS) more than 6 months ago. This may include procedures that do not involve the conjunctiva such as Hydrus Microstent, iStent and endoscopic cyclophotocoagulation (ECP) laser.

The authors do not think it likely that pseudophakia will influence the outcomes but randomisation will be stratified by lens status to ensure balance in the treatment arms.

Exclusion Criteria:

General Exclusion Criteria

Patients are ineligible to participate in the study where any of the following criteria apply:

* Any inclusion criteria not met.
* Pregnant or nursing women (or planning pregnancy).
* Unwilling or unable to give informed consent, unwilling to accept randomisation, or unable to return for scheduled protocol visits.
* Ongoing participation in other interventional clinical trials. Exclusion criteria for study eye

The patient may not be entered into the study if any of the following exclusion criteria are present in the study eye:

* No light perception vision.
* Active diabetic retinopathy.
* Secondary glaucomas.
* Unwilling to discontinue contact lens use after surgery.
* Conjunctival scarring from prior ocular trauma or cicatrizing disease (e.g. Stevens Johnson syndrome, ocular pemphigoid) precluding a superior trabeculectomy.
* Functionally significant cataract likely to require surgery within 6 months of glaucoma surgery.
* Previous complicated cataract surgery in the study eye.
* Need for glaucoma surgery combined with other ocular procedures (i.e. cataract surgery, penetrating keratoplasty, or retinal surgery) or anticipated need for additional ocular surgery.
* Iris neovascularization or proliferative retinopathy.
* Iridocorneal endothelial syndrome.
* Epithelial or fibrous downgrowth.
* Chronic or recurrent uveitis.
* Steroid-induced glaucoma.
* Severe posterior blepharitis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate: | 6 months
  The number of potential participants enrolled over a set time

SECONDARY OUTCOMES:
Success rate | 6 months
  Eyes that have not failed and are not on supplemental medical therapy are considered complete successes
Failure rate | 6 months
  * IOP >21 mmHg or not reduced by 20% below baseline on two consecutive follow-up visits
  * Additional glaucoma surgery
  * Loss of vision.
  * IOP <5 mmHg on two consecutive follow-up visits
Complication rate | 6 months
The number of extra unscheduled clinic visits and unplanned procedures | 6 months
Loss to follow-up rate | 6 months
Response rates to the self-report | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: K Sheng Lim, MD, Principal Investigator — Guy's and St Thomas NHS Foundation Trust
Locations (1):
- St Thomas Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No